CLINICAL TRIAL: NCT02636725
Title: A Phase II Trial of Concurrent Axitinib and Pembrolizumab in Subjects With Advanced Alveolar Soft Part Sarcoma (ASPS) and Other Soft Tissue Sarcomas (STS)
Brief Title: Axitinib and Pembrolizumab in Subjects With Advanced Alveolar Soft Part Sarcoma and Other Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonathan Trent, MD, PhD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Trent, MD, PhD, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150932
Record Dates: First submitted 2015-12-14; First posted 2015-12-22 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Alveolar Soft Part Sarcoma; Soft Tissue Sarcomas
Keywords: Advanced Alveolar Soft Part Sarcoma; ASPS; STS
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Sarcoma | interventions — Axitinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axitinib Plus Pembrolizumab Group (Experimental): Participants in this group will receive combination treatment of Axitinib plus Pembrolizumab for up to 2 years followed by monotherapy of Axitinib until withdrawal of consent, disease progression and/or unacceptable toxicity as assessed by treating physician, whichever occurs first.
  Interventions: Drug: Axitinib; Drug: Pembrolizumab
- Axitinib Plus Pembrolizumab Expansion Cohort (Experimental): Expansion cohort for up to 10 additional patients with alveolar soft part sarcoma. Participants in this group will receive combination treatment of Axitinib plus Pembrolizumab for up to 2 years followed by monotherapy of Axitinib until withdrawal of consent, disease progression and/or unacceptable toxicity as assessed by treating physician, whichever occurs first.
  Interventions: Drug: Axitinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Axitinib — 5 mg tablets twice daily oral dose administered for 7 consecutive weeks on Cycle 1. A safety lead-in consisting of the initial five patients, intrapatient dose escalation of Axitinib will be permitted based on the absence of predefined toxicities. Twice daily oral dose between 2 mg to 10 mg Axitinib tablets will be administered on subsequent 6 week cycles until withdrawal of consent, disease progression and/or unacceptable toxicity as assessed by treating physician, whichever occurs first.
  Other Names: Inlyta
Drug: Pembrolizumab — 200 mg intravenous infusion administered every 21 weeks beginning week 2 of Cycle 1 for a maximum of up to 2 years or until withdrawal of consent, disease progression and/or unacceptable toxicity as assessed by treating physician, whichever occurs first.
  Other Names: MK-3475; Keytruda

SUMMARY:
The purpose of this research study is to test if Axitinib together with Pembrolizumab can slow tumor growth and know the side effects of the combination treatment.

DETAILED DESCRIPTION:
Arm 2, the Axitinib Plus Pembrolizumab Expansion Cohort, did not open.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed sarcoma with pathology review required for any outside samples.
2. The following histologies may be enrolled without prior treatment:

   * alveolar soft part sarcoma,
   * clear cell sarcoma,
   * epithelioid hemangioendothelioma, and
   * chordoma.
3. The following histologies may be enrolled only if refractory to anthracycline-based chemotherapy or if the patient refuses to undergo standard of care treatment:

   * synovial sarcoma,
   * rhabdomyosarcoma,
   * malignant peripheral nerve sheath tumors,
   * dedifferentiated, pleomorphic or myxoid/round cell liposarcoma,
   * leiomyosarcoma,
   * malignant phylloides tumor,
   * high grade undifferentiated pleomorphic sarcomas (HGUPS/MFH),
   * angiosarcoma,
   * spindle cell sarcoma, not otherwise specified (NOS)
   * malignant myoepithelioma.
4. The following histologies may be enrolled only if refractory to at least one line of chemotherapy or if the patient refuses to undergo standard of care treatment:

   * solitary fibrous tumor/hemangiopericytoma.
5. The following histologies may be enrolled only if refractory to at least first-line targeted therapy or if the patient refuses to undergo standard of care treatment:

   * gastrointestinal stromal tumors,
   * extraskeletal myxoid chondrosarcoma,
   * PEComa.
6. Primary tumors of bone including Ewing's sarcoma, osteosarcoma, and dedifferentiated chondrosarcoma may only be enrolled if there are measurable target lesions occurring in soft tissue and they are refractory to standard of care anthracycline-based chemotherapy.
7. Any other histology or standard of care therapy not specifically addressed will be reviewed by the principal investigator and pathologist for final determination of eligibility.
8. Measurable disease as defined by RECIST v1.1.
9. Radiographic progression as defined by RECIST v1.1, based on comparison between two radiographic studies no greater than 6 months apart.
10. Inability to undergo complete resection of the disease by surgery.
11. Adequate organ function as defined:

    * Hematological

      * Absolute neutrophil count (ANC) ≥1,000 / microliter (mcL)
      * Platelets ≥75,000 / mcL
      * Hemoglobin ≥8 g/dL without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
    * Renal

      * Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN. (GFR can also be used in place of creatinine or CrCl). Creatinine clearance should be calculated per institutional standard.
    * Hepatic

      * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN.
      * Aspartate Aminotransferase (AST/SGOT) and Alanine Transaminase (ALT/SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases.
      * Albumin >2.5 mg/dL
    * Coagulation

      * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
      * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
12. Age ≥ 16 years.
13. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
14. Patients must consent and be willing to undergo three core needle biopsies at baseline, prior to starting Cycle 3, and at off-study. At least one tumor site must be amenable to biopsy in the judgment of the interventional radiologist.
15. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
16. Females of child bearing potential that are sexually active must agree to either practice 2 medically accepted highly effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 120 days after the last dose of study drug. See Appendix G for protocol-approved highly effective methods of contraceptive combinations. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    * Negative test for pregnancy is required of females of child-bearing potential; A female of child bearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1. has not undergone a hysterectomy or bilateral oophorectomy; or 2. has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months or 730 days).
    * Conception while on treatment must be avoided
17. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Prior history of vasectomy does NOT replace requirement for contraceptive use.
18. Suitable venous access to allow for all study related blood sampling
19. Ability to understand and willingness to sign a written informed consent document.
20. For minors that are 16 to 18 years of age, assent and parental (or legally acceptable representative) written informed consent must be obtained.

Exclusion Criteria:

1. Prior therapy with axitinib. Patients are permitted to have received prior tyrosine kinase inhibitor (TKI) therapy including imatinib, sunitinib, pazopanib, or similar. Patients may have received prior Programmed death 1 (PD-1)/Programmed death-ligand 1 (PD-L1) directed therapy.
2. Hypersensitivity to axitinib, pembrolizumab or any of its excipients.
3. Patients may not be receiving any other investigational agents (within 4 weeks prior to Cycle 1, day 1).
4. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Cycle 1, day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Patient has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle 1, Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Additional known malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
7. Patients with end-organ dysfunction as defined in inclusion criterion (i.e. #11 above).
8. Patients with bone-only lesions.
9. Patients with underlying immune deficiency, chronic infections including HIV, hepatitis, or tuberculosis (TB) or autoimmune disease.
10. Patients with underlying hematologic issues including bleeding diathesis, known previous GI bleeding requiring intervention within the past 6 months, active pulmonary emboli or deep vein thromboses (DVT) that are not stable on anticoagulation regimen.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Concomitant (or receipt of) treatment with medications that may affect the metabolism of pembrolizumab and/or axitinib within 7 days prior to Cycle 1, day 1 of axitinib.
14. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
17. Prolonged corrected QT (QTc) interval on Screening EKG >475 ms.
18. Ejection Fraction <40% by 2D echocardiogram (ECHO) at Screening.
19. Any serious medical or psychiatric illness/condition including substance use disorders likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.
20. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Trent, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilky BA, Trucco MM, Subhawong TK, Florou V, Park W, Kwon D, Wieder ED, Kolonias D, Rosenberg AE, Kerr DA, Sfakianaki E, Foley M, Merchan JR, Komanduri KV, Trent JC. Axitinib plus pembrolizumab in patients with advanced sarcomas including alveolar soft-part sarcoma: a single-centre, single-arm, phase 2 trial. Lancet Oncol. 2019 Jun;20(6):837-848. doi: 10.1016/S1470-2045(19)30153-6. Epub 2019 May 8. PMID 31078463

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axitinib Plus Pembrolizumab Group
Started | 33
Completed | 32
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib Plus Pembrolizumab Group
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 24
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 29
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Evaluable Participants Achieving Progression-Free Survival (PFS) at 3 Months
Description: Percentage of participants who are disease progression free 3 months after initiation of therapy. Disease progression will be evaluated from imaging measures using the Response Evaluation Criteria for Solid Tumors (RECIST) 1.1.
Time Frame: 3 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib Plus Pembrolizumab Group
Number analyzed (Participants) | 33
percentage of participants | 81.8 [63.9 to 91.4]

2. Secondary Outcome: Percentage of Evaluable Participants Achieving Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as achieving complete response (CR) or partial response (PR) from imaging measures using (RECIST) 1.1.
Time Frame: Up to 2 Years
Population: Evaluable participants received at least 80% of scheduled axitinib doses and two infusions of pembrolizumab, have measurable disease at baseline and at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib Plus Pembrolizumab Group
Number analyzed (Participants) | 32
percentage of participants | 28.1 [13.8 to 46.8]

3. Secondary Outcome: Percentage of Evaluable Participants Achieving Clinical Benefit Response (CBR)
Description: CBR is defined as achieving complete response (CR), partial response (PR) or stable disease (SD) from imaging measures using (RECIST) 1.1.
Time Frame: Up to 2 Years
Population: Participants that received at least 80% of scheduled axitinib doses and two infusions of pembrolizumab, have measurable disease at baseline and at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib Plus Pembrolizumab Group
Number analyzed (Participants) | 32
percentage of participants | 59.4 [40.6 to 76.3]

4. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) is defined as time from treatment initiation until documented disease progression according to Response Evaluation Criteria for Solid Tumors version 1.1 (RECIST v1.1) or death (by any cause, in the absence of progression). In progression-free patients, PFS will be censored at the last evaluable tumor assessment.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib Plus Pembrolizumab Group
Number analyzed (Participants) | 33
months | 9.3 [3.7 to 12.3]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is (OS) is defined as the time from treatment initiation to death from any cause, whichever is earlier. Participants alive or those lost to follow-up will be censored at the last date of contact (or last date known to be alive).
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib Plus Pembrolizumab Group
Number analyzed (Participants) | 33
months | 18.7 [12.4 to 58.4]

6. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs), Dose-Limiting Toxicities, and Grade 3 or Higher Treatment-Emergent Adverse Events
Description: The number of participants experiencing serious adverse events (SAEs), dose-limiting toxicities (DLTs), and grade 3 or higher treatment-emergent adverse events (AEs). AEs, SAEs and DLTs will be evaluated by treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03. Treatment-emergent adverse events are those found to be definitely, probably and possibly related to study therapy.
Time Frame: Up to 25 months
Measure: Number; unit: participants
Arm/Group | Axitinib Plus Pembrolizumab Group
Number analyzed (Participants) | 33
participants
  Serious Adverse Events (SAEs) | 9
  Dose Limiting Toxicities (DLTs) | 7
  Grade 3 or higher treatment-emergent AE (excluding SAE and DLT) | 6

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Axitinib Plus Pembrolizumab Group
All-Cause Mortality (participants affected / at risk) | 22/33
Serious Adverse Events (participants affected / at risk) | 9/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib Plus Pembrolizumab Group (N=33)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Nausea and Vomiting
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Investigations - Other (Investigations) | 1 (1) — Transaminitis
Papulopustular rash (Infections and infestations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Radiculitis (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) — Acute renal failure
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) — Uremia
Seizure (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib Plus Pembrolizumab Group (N=33)
Abdominal Pain (Gastrointestinal disorders) | 12 (20)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 14 (26)
Alkaline phosphatase increased (Investigations) | 10 (16)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (8)
Anorexia (Metabolism and nutrition disorders) | 12 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 13 (23)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Bloating (Gastrointestinal disorders) | 2 (5)
Blood bilirubin increased (Investigations) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest Pain - Cardiac (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (22)
Creatinine increased (Investigations) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 26 (53)
Dry Mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 4 (4) — Ear congestion
Ear Pain (Ear and labyrinth disorders) | 2 (2)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 26 (56)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (8)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Acid reflux
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (3) — Mouth sensitivity
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Mouth soreness
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Rectal irritation
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Stomatitis
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Decreased appetite
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Headaches (morning)
General disorders and administration site conditions - Other (General disorders) | 1 (2) — Itching skin
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Weakness
Headache (Nervous system disorders) | 5 (11)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemoglobin increased (Investigations) | 5 (7)
Hemorrhoids (Gastrointestinal disorders) | 3 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hypertension (Vascular disorders) | 14 (21)
Hyperthyroidism (Endocrine disorders) | 2 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 18 (18)
Immune system disorders - Other (Immune system disorders) | 1 (1) — Disseminated Herpes Zoster
Infections and infestations - Other (Infections and infestations) | 1 (1) — Herpes simplex - Eye lesion
Insomnia (Psychiatric disorders) | 5 (5)
Investigations - Other (Investigations) | 1 (1) — Elevated triglycerides
Investigations - Other (Investigations) | 3 (3) — Elevated thyroid stimulating hormone (TSH)
Investigations - Other (Investigations) | 1 (1) — Eosinophilia
Investigations - Other (Investigations) | 2 (2) — Hand sensitivity
Investigations - Other (Investigations) | 1 (1) — Hyperlipidemia
Investigations - Other (Investigations) | 1 (2) — Increased blood urea nitrogen (BUN)
Investigations - Other (Investigations) | 1 (1) — Lung discomfort
Investigations - Other (Investigations) | 1 (1) — Mouth sensitivity
Investigations - Other (Investigations) | 1 (1) — Mouth sensitivity - spicy foods
Investigations - Other (Investigations) | 1 (2) — Mouth sores
Investigations - Other (Investigations) | 1 (1) — Muscle aches
Investigations - Other (Investigations) | 1 (1) — Sputum production
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (3)
Mucositis Oral (Gastrointestinal disorders) | 14 (27)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Foot sensitivity
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (2) — Hand sensitivity
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Intermittent hand sensitivity
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Oligoarthritis
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 19 (33)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Hand sensitivity
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Right-sided sciatica
Non-cardiac chest pain (General disorders) | 5 (6)
Oral dysesthesia (Gastrointestinal disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2)
Oral Pain (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 17 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (11)
Papulopustular rash (Infections and infestations) | 8 (9)
Paresthesia (Nervous system disorders) | 3 (4)
Platelet count decreased (Investigations) | 3 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) — Urinary urgency
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) — Glycosuria
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2 (3) — Vaginal irritation
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hemoptysis
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Rhinorrhea
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Shortness of breath with exertion
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Acne
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Eczema exacerbation
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Fingertip sensitivity
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Foot rash
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2) — Foot sensitivity
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Hand and foot sensitivity
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Lip skin thickening
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Skin irritation
Stomach pain (Gastrointestinal disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 4 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (19)
Weight loss (Investigations) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
White blood cell decreased (Investigations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Tooth Infection (Infections and infestations) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Skin lesions
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Hand nodules
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Left scalp lesion
Sinus tachycardia (Cardiac disorders) | 2 (4)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Nose dryness
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Post-viral bronchitis
Reproductive system and breast disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (3) — Herpes simplex virus (HSV) Flare
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) — Acute renal insufficiency
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) — Mood changes
Presyncope (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Right leg neuropathy
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Right arm neuropathy
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Altered mental status
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Right neck pulsation
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Shoulder dislocation
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Right ankle sprain
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Intermittent muscle spasms
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) — Hyponatremia
Investigations - Other (Investigations) | 1 (1) — Left Chest pressure/sharpness with inspiration
Investigations - Other (Investigations) | 1 (1) — Lower respiratory infection
Investigations - Other (Investigations) | 1 (1) — Soreness and bruising at biopsy site
Investigations - Other (Investigations) | 1 (1) — Tooth Abcess
Investigations - Other (Investigations) | 1 (1) — Tooth pain
Investigations - Other (Investigations) | 1 (1) — Cold like symptoms
Infections and infestations - Other (Infections and infestations) | 1 (1) — Not otherwise specified (NOS)
Infections and infestations - Other (Infections and infestations) | 1 (1) — Fungal groin infection
Infections and infestations - Other (Infections and infestations) | 1 (1) — Upper respiratory infection with low grade fever
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Cold
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Diaphragm cramping intermittent
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Diffuse body aches
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Dysuria
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Fainting
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Neck pain
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Night sweats
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Right Inner Thigh Muscular Pain with Noticeable Tumor Inflammation
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Runny nose
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Tongue sensitity
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2) — Thrush
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Flu like symptoms (General disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1) — Thrombocytopenia
Atrial fibrillation (Cardiac disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Arm 2, the Axitinib Plus Pembrolizumab Expansion Cohort, did not open.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT02636725/Prot_SAP_000.pdf